CLINICAL TRIAL: NCT06210880
Title: Change of Gastric Fluid Volume After Oral Hydration in Fasted Objects
Status: Not yet recruiting | Type: Observational
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Professor, SMG-SNU Boramae Medical Center
Other Study IDs: 10-2023-32
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Preoperative Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the permissive amount and time limit of clear fluid intake for preoperative fasting.

DETAILED DESCRIPTION:
Observations of two kinds of liquids (water, carbohydrate drink) in five different volumes (10ml, 50ml, 100ml, 200ml, 400ml) will be performed on different days. Subjects prepare for investigation, a 4-hour fast excluding water, followed by 1 hour of fasting including water, and then 10 ml or 50 ml or 100 ml or 200 ml or 400 ml of clear water in a pre-randomized order and then the cross-sectional area of the stomach antrum will be measured via ultrasound every 10-minute until the contents are no longer visible. The same observation will be performed with a noNPO drink beverage containing 50 g of carbohydrate, again in a randomized order, and then 10 ml, 50 ml, 100 ml, 200 ml or 400 ml, and then every 10 minutes until the contents are no longer visible. One dose of one type of fluid will be ingested and observed at each visit, and repeated visits will be made until observations for all doses have been completed (10 visits in total, with 5 doses of water and carbohydrate drinks). During measurement, the stomach will be checked for contents supine position and then turned to the right decubitus.

ELIGIBILITY:
Inclusion Criteria:

* age ≥19 yrs

Exclusion Criteria:

* history of abdominal surgery

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers over 19 years old without a history of abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-02-22 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
gastric volume | 10 min
  measure by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Young Hwang, MD,PhD, Study Chair — SMG-SNU Boramae Medical Center
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Warner MA, Warner ME, Weber JG. Clinical significance of pulmonary aspiration during the perioperative period. Anesthesiology. 1993 Jan;78(1):56-62. doi: 10.1097/00000542-199301000-00010. PMID 8424572
- [Background] Lienhart A, Auroy Y, Pequignot F, Benhamou D, Warszawski J, Bovet M, Jougla E. Survey of anesthesia-related mortality in France. Anesthesiology. 2006 Dec;105(6):1087-97. doi: 10.1097/00000542-200612000-00008. PMID 17122571
- [Background] Neelakanta G, Chikyarappa A. A review of patients with pulmonary aspiration of gastric contents during anesthesia reported to the Departmental Quality Assurance Committee. J Clin Anesth. 2006 Mar;18(2):102-7. doi: 10.1016/j.jclinane.2005.07.002. PMID 16563326
- [Background] Bolondi L, Bortolotti M, Santi V, Calletti T, Gaiani S, Labo G. Measurement of gastric emptying time by real-time ultrasonography. Gastroenterology. 1985 Oct;89(4):752-9. doi: 10.1016/0016-5085(85)90569-4. PMID 3896910
- [Background] Milling TJ Jr, Rose J, Briggs WM, Birkhahn R, Gaeta TJ, Bove JJ, Melniker LA. Randomized, controlled clinical trial of point-of-care limited ultrasonography assistance of central venous cannulation: the Third Sonography Outcomes Assessment Program (SOAP-3) Trial. Crit Care Med. 2005 Aug;33(8):1764-9. doi: 10.1097/01.ccm.0000171533.92856.e5. PMID 16096454